CLINICAL TRIAL: NCT00384111
Title: A Phase 3 Open Label Multicenter, Randomized Study to Compare the Efficacy and Safety of the Zevalin (Ibritumomab Tiuxetan) Therapeutic Regimen Following Cyclophosphamide, Vincristine, Prednisone, and Rituximab (R-CVP) With R-CVP Alone in High-Risk Subjects With Previously Untreated CD20-Positive Follicular Non-Hodgkin's Lymphoma
Brief Title: Phase 3 Study of Zevalin Following R-CVP in Previously Untreated Patients With Follicular Non Hodgkin's Lymphoma (NHL)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated early as per the Sponsor's decision.
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Collaborators: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 106NH301
Record Dates: First submitted 2006-10-03; First posted 2006-10-05 (Estimated); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Follicular Lymphoma; Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive standard R-CVP followed by Zevalin Therapeutic Regimen (Day 1: 250 mg/m2 Rituxan followed by 5 mCi 111In Zevalin Day 7: 250 mg/m2 Rituxan followed by 0.4 mCi/kg Zevalin).
  Interventions: Drug: Zevalin Therapeutic Regimen; Drug: R-CVP
- 2 (Active Comparator): Participants will receive standard R-CVP.
  Interventions: Drug: R-CVP

INTERVENTIONS:
Drug: Zevalin Therapeutic Regimen — Day 1: 250 mg/m2 Rituxan followed by 5 mCi 111In Zevalin. Day 7: 250 mg/m2 Rituxan followed by 0.4 mCi/kg Zevalin
  Arms: 1
Drug: R-CVP — Standard R-CVP

SUMMARY:
This study will treat follicular lymphoma patients who have not received previous treatment with R-CVP. Half of the patients will receive Zevalin after R-CVP and the other half will receive only R-CVP. The two patient groups will be compared to determine if Zevalin given after R-CVP therapy provides greater benefits than receiving no additional anti-cancer therapy after R-CVP.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent and any authorizations required by local law (e.g., Protected Health Information).
* Age greater than or equal to 18 years at the time of informed consent.
* Histologically confirmed follicular NHL according to the Revised European American Lymphoma (REAL)/World Health Organization (WHO)classification (from initial diagnosis); grades 1, 2, or 3.
* Bi-dimensionally measurable lesion(s) in at least one site.
* High risk NHL as defined by a follicular lymphoma international prognostic index (FLIPI) of 3, 4, or 5 assessed within 3 months prior to randomization.
* NHL requires treatment as determined by the investigator.
* Confirmed CD20+ lymphoma cells.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1,or 2.
* Expected survival of greater than or equal to 3 months.
* Male subjects and female subjects of child bearing potential willing to practice effective contraception during the study and willing and able to continue contraception for 1 year after their last dose of study treatment (R CVP for subjects in the observation arm and the Zevalin therapeutic regimen for subjects in the Zevalin arm).

Exclusion Criteria:

* Previous anticancer treatment for NHL, including chemotherapy, immunotherapy, radiation (locoregional or extended field), radioimmunotherapy, or investigational therapy.
* Known seropositivity for hepatitis C virus, hepatitis B virus (surface antigen-positive), or other active infection uncontrolled by treatment.
* Known diagnosis of human immunodeficiency virus infection.
* Presence of primary gastric, central nervous system (CNS), or testicular lymphoma, or transformed lymphoma, or chronic lymphocytic leukemia (CLL).
* Active therapy within previous 5 years for other malignancy, except non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma.
* Abnormal liver function: total bilirubin >1.5 X upper limit of normal (ULN) or ALT >2.5 X ULN.
* Impairment of renal function (serum creatinine >1.5 X ULN) not due to lymphoma.
* Concurrent severe and/or uncontrolled medical disease (e.g., uncontrolled diabetes, congestive heart failure, myocardial infarction within 6 months of study, unstable and uncontrolled hypertension, chronic renal disease, or active uncontrolled infection) that could compromise participation in the study.
* Known hypersensitivity to murine and/or chimeric proteins.
* History of severe allergic or anaphylactic reactions.
* Known allergy to any components present in rituximab, cyclophosphamide, vincristine, and prednisone (CVP), or Zevalin.
* Treatment with another study treatment or approved therapy for investigational use within the 12 weeks prior to randomization.
* Exposure to monoclonal antibodies, cytokines, growth factors, soluble receptors, other recombinant products, or fusion proteins.
* Females with a positive pregnancy test result at screening or who are currently breastfeeding.
* Inability to comply with study requirements.
* Major surgery within 28 days except for diagnosis.
* In need of immediate intervention to treat life threatening complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Gulfcoast Oncology Associates, St. Petersburg, Florida
  - Wellstar-Northwest Georgia Oncology Centers, Marietta, Georgia
  - Oncology Hematology Care Inc., Cincinnati, Ohio
  - Chattanooga Oncology Hematology Care, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: It was planned to randomized the enrolled subjects to receive R-CVP followed by Zevalin Therapeutic Regimen or R-CVP. However, due to low enrollment and early termination, participants were not randomized and received any treatment. The data for the Participant flow and Baseline sections is reported for all enrolled participants in one arm.
Groups:
- All Enrolled Participants: Participants with follicular lymphoma who have not received previous treatment with R-CVP were enrolled in the study.
Period: Overall Study
Arm/Group | All Enrolled Participants
Started | 26
Completed | 0
Not Completed | 26
Not completed — Disease Progression | 3
Not completed — Adverse Event | 1
Not completed — Investigator Decision | 3
Not completed — Study Terminated by the Sponsor | 19

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: 18 months
Population: Data for this outcome measure was not collected and summarized as the study was terminated early by the sponsor.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Time Frame: 18 months
Population: Data for this outcome measure was not collected and summarized as the study was terminated early by the sponsor.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to end of study (approximately up to 4 years)
Description: Safety data were not collected as the study was terminated early by the sponsor.
Arm/Group | All Enrolled Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Outcome measures and safety data were not collected and summarized as the study was terminated early by the sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No